CLINICAL TRIAL: NCT03115268
Title: Delivering Group Support for People With Aphasia Through Eva Park
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City, University of London (Other)
Collaborators: The Stroke Association, United Kingdom (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: TSA 2016/05
Record Dates: First submitted 2017-03-24; First posted 2017-04-14 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2018-07

CONDITIONS: Aphasia
Keywords: social support
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate (Experimental): Participants allocated to the immediate arm will receive 6 months of Social support groups delivered in EVA Park immediately after randomisation. They will be re-assessed in Month 7, then receive 6 months of usual care, followed by reassessment in month 14.
  Interventions: Behavioral: Social support groups delivered in EVA Park
- Wait list control (Active Comparator): Participants allocated to the wait list control arm will receive 6 months of usual care after randomisation. They will be re-assessed in month 7, and will then receive 6 months of social support groups delivered in EVA Park, with reassessment in month 14.
  Interventions: Behavioral: Social support groups delivered in EVA Park

INTERVENTIONS:
Behavioral: Social support groups delivered in EVA Park — Intervention will comprise support group meetings delivered in EVA Park, a virtual island created for people with aphasia. Scheduled meetings will be held every two weeks, led by the group co-ordinator and volunteers. Participants will have unlimited access to EVA Park, so will be able to meet up with other group members between meetings.

SUMMARY:
The project will investigate the feasibility and acceptability of a remote support group intervention for people with aphasia, and will investigate the impact of that intervention on measures of wellbeing, quality of life and communication. The intervention will be delivered to 32 participants in Eva Park, a virtual island specifically designed for people with aphasia.

ELIGIBILITY:
Inclusion Criteria:

* Stroke survivor with aphasia; Score within the aphasic range on the Frenchay Aphasia Screening Test (FAST); Fluent pre-stroke user of English.

Exclusion Criteria:

* Co-morbidity affecting cognition; Severe hearing or visual impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Pre to post intervention change on the Warwick Edinburgh Mental Well-being Scale (WEMWBS) | At randomisation and at 7 and 14 months post randomisation
  A 14 item questionnaire about feelings of wellbeing
Pre to post intervention change on the Communication Activities of Daily Living test (CADL-2) | At randomisation and at 7 and 14 months post randomisation
  A 50 item standardized test of everyday communication activities, designed for people with aphasia

SECONDARY OUTCOMES:
Pre to post intervention change on the Social Connectedness Scale - Revised (Lee et al. 2001) | At randomisation and at 7 and 14 months post randomisation
  A 20 item questionnaire about feelings of social connectedness
Pre to post intervention change on The Western Aphasia Battery - Revised (Kertesz, 2007) | At randomisation and at 7 and 14 months post randomisation
  A standardized assessment of language impairment designed for people with aphasia
Pre to post intervention change on the Stroke and Aphasia Quality of Life measure (SAQOL-39) (Hilari et al, 2003) | At randomisation and at 7 and 14 months post randomisation
  A self reporting questionnaire about health related quality of life designed for people with stroke and aphasia

OTHER OUTCOMES:
Participant recruitment and attrition rates | Throughout recruitment, intervention and follow up period, up to 14 months
  The number of participants referred to the project and the proportion who consent; the number of individuals lost to follow up
Participant views about intervention | Interviews conducted up to 4 weeks post intervention (Month 7 for immediate arm; month 14 for waitlist control arm)
  Responses to in-depth semi-structured interviews conducted with all participants post intervention
Group coordinators' and volunteers' views about intervention | At month 7 for the immediate arm; at month 14 for the waitlist control arm
  Responses to in-depth semi-structured interviews conducted with all coordinators and 8 purposefully selected volunteers
Qualitative findings from Human Computer Interaction Assessments | Conducted in the first and last week of intervention; Months 1 and 6 for the immediate arm; Months 8 and 13 for the waitlist control arm.
  Structured observations and interviews conducted with 8 randomly selected participants from each arm, aiming to determine the suitability of EVA Park for delivering support group meetings
Time spent using EVA Park | throughout intervention periods; Months 1 - 6 for the immediate arm; Months 8 - 13 for the waitlist control arm
  Automatic log data of each participant's usage of EVA Park
Treatment cost | Throughout intervention periods; Months 1 - 6 for the immediate arm; Months 8 - 13 for the waitlist control arm.
  Logs of all costs associated with the intervention, relating to: Human Resources, Technical costs, Materials, Capital costs and Travel

CONTACTS AND LOCATIONS:
Overall Officials: Jane Marshall, PhD, Principal Investigator — City, University of London
Locations (1):
- City, University of London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Marshall J, Devane N, Talbot R, Caute A, Cruice M, Hilari K, MacKenzie G, Maguire K, Patel A, Roper A, Wilson S. A randomised trial of social support group intervention for people with aphasia: A Novel application of virtual reality. PLoS One. 2020 Sep 24;15(9):e0239715. doi: 10.1371/journal.pone.0239715. eCollection 2020. PMID 32970784